CLINICAL TRIAL: NCT04744922
Title: Clinical and Biological Effects of Citrus-phytochemicals in Subjective Cognitive Decline: a Pilot Randomized Controlled Trial.
Brief Title: Clinical and Biological Effects of Citrus-phytochemicals in Subjective Cognitive Decline.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: University of Chieti (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 270/2020
Record Dates: First submitted 2021-02-05; First posted 2021-02-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-03

CONDITIONS: Subjective Cognitive Decline
Keywords: Citrus-phytochemicals, auraptene, naringenin; subjective cognitive decline, randomized, efficacy; cognitive tests, R-BANS, interleukins, Interleukin-8

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auraptene and Naringenin Arm (Experimental): One capsule a day for 9 months
  Interventions: Dietary Supplement: Extracts of citrus peels standardized in AUR and NAR (phytocomplex).
- Control Arm (Placebo Comparator): One capsule a day for 9 months
  Interventions: Dietary Supplement: Extracts of citrus peels standardized in AUR and NAR (phytocomplex).

INTERVENTIONS:
Dietary Supplement: Extracts of citrus peels standardized in AUR and NAR (phytocomplex). — One capsule a day for 9 months

SUMMARY:
Subjective cognitive decline (SCD) is receiving increasing attention as a risk factor for incident dementia due to AD. SCD manifests prior to the onset of clinical impairment, and as such could serve as a potential target population for early intervention trials. The pathogenesis of AD is complex and involves a dysregulation of the neuroendocrine immune (NEI) system, a network of signaling molecules, such as neurotransmitters, hormones and cytokines. As a result, it may be unlikely that cognitive decline may be mitigated by drugs acting on a single specific target. Plant extracts acting at different levels of the NEI regulation could represent appealing therapeutic strategies for cognitive decline. Citrus-derived phytochemicals, like auraptene and naringenin, showed antioxidant, anti-inflammatory, and neuroprotective effects in preclinical studies of AD mouse models and preservation of cognition in elderly without cognitive impairment. This is a pilot randomized controlled trial to determine clinical and biological effects of Citrus-phytochemicals in individuals with SCD. Participants will be randomized to receive Citrus-phytochemicals standardized in auraptene and naringenin or placebo for 9 months. Cognitive tests and blood-based biological markers will be done at baseline and at the end of treatment as outcome measures.

DETAILED DESCRIPTION:
Background: Alzheimer's disease (AD) is a neurodegenerative disorder which represents a major health issue and financial burden for health care systems around the world. The impact will further increase over the next decades due to increasing life expectancies. AD leads to progressive and irreversible disturbances of cognition and functional abilities. AD is the fifth-leading cause of death among those age 65 and older and is also a leading cause of disability and poor health. Due to the absence of a cure against AD, the public health priority has focused more recently on improvement of cognitive performance in older age and, possibly, prevention of cognitive decline. Subjective cognitive decline (SCD) in older adults is increasingly recognized as a potential indicator of non-normative cognitive decline and eventual progression to dementia. Longitudinal studies in SCD showed an up to 4.5-fold increased risk for progression to mild cognitive impairment. SCD has also been characterized by pathological changes of the brain associated with AD. These findings suggest that SCD may be an early clinical marker for AD, making an ideal target to test preventive interventions. Several nutraceuticals have displayed over the years the ability or potential to improve cognitive impairment. Among these, auraptene (AUR) and naringenin (NAR) are natural bioactive compounds derived from peels of Citrus fruits, with a strong preclinical rationale for cognitive enhancement. In fact, preclinical studies showed that they have anti-inflammatory, antioxidant, and neuroprotective effects in mouse brain and, specifically, in AD mouse models. These effects are mediated by a number of neuropeptides, growth factors, hormones, and cytokines, which are components of the neuroendocrine and immune (NEI) system, a complex network of communication, which showed altered functioning in ageing and neurodegenerative diseases.

The capacity of some nutraceutical in restoring and remodelling the NEI response at both neuroendocrine and immune level, could represent a new strategy in order to reach healthy ageing and prevent cognitive decline in the elderly. This perspective is supported by the results of a randomized, placebo-controlled, double blind study of 84 older adults, in which administration of AUR for 24 weeks showed significantly higher percentage of improvement in the immediate memory in the AUR group compared to the placebo.

Specific aims: This is a pilot randomized controlled trial to determine the cognitive and biological effects of Citrus peels extracts standardized in auraptene and naringenin, in individuals with SCD.

Specific aim 1. The investigators will enrol 80 individuals with SCD randomized into two groups of treatments, i.e. control and Citrus peels extracts. Cognitive assessment will be carried out at baseline and after 9 months of treatment, in order to evaluate the effect on cognition.

The investigators hypothesize that treatment group has an improvement in cognition compared to placebo group.

Specific aim 2. To evaluate the biological effects of the Citrus peels extracts treatment on the NEI system, through blood samples taken at baseline, and after 9 months of treatment.

The investigators hypothesize that treatment group has an improvement in the NEI functions as indicated by biological markers (increase of the growth factors, reduction of stress hormones levels, reduction of inflammation) compared to placebo group.

ELIGIBILITY:
Inclusion Criteria:

* subjective cognitive decline,
* lack of objective cognitive impairment.

Exclusion Criteria:

* clinically significant depression and anxiety,
* psychiatric disorders,
* unstable medical conditions.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Cognitive outcome | 9 months
  Repeatable Battery for the Assessment of the Neuropsychological Status (R-BANS).
  The minimum score is 40 and the maximum is 160. Higher scores mean a better performances.

SECONDARY OUTCOMES:
Biological outcome | 9 months
  Interleukin-8

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Galluzzi, Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data collected in this study will not be publicly available but will be provided to any qualified researcher interested in the topic of this project, upon presentation of a research study and approval of the local Ethics Committee.
Access Criteria: Local Ethics Committee approval.

REFERENCES:
- [Background] Rebello CJ, Beyl RA, Lertora JJL, Greenway FL, Ravussin E, Ribnicky DM, Poulev A, Kennedy BJ, Castro HF, Campagna SR, Coulter AA, Redman LM. Safety and pharmacokinetics of naringenin: A randomized, controlled, single-ascending-dose clinical trial. Diabetes Obes Metab. 2020 Jan;22(1):91-98. doi: 10.1111/dom.13868. Epub 2019 Sep 30. PMID 31468636
- [Background] Jessen F, Amariglio RE, van Boxtel M, Breteler M, Ceccaldi M, Chetelat G, Dubois B, Dufouil C, Ellis KA, van der Flier WM, Glodzik L, van Harten AC, de Leon MJ, McHugh P, Mielke MM, Molinuevo JL, Mosconi L, Osorio RS, Perrotin A, Petersen RC, Rabin LA, Rami L, Reisberg B, Rentz DM, Sachdev PS, de la Sayette V, Saykin AJ, Scheltens P, Shulman MB, Slavin MJ, Sperling RA, Stewart R, Uspenskaya O, Vellas B, Visser PJ, Wagner M; Subjective Cognitive Decline Initiative (SCD-I) Working Group. A conceptual framework for research on subjective cognitive decline in preclinical Alzheimer's disease. Alzheimers Dement. 2014 Nov;10(6):844-52. doi: 10.1016/j.jalz.2014.01.001. Epub 2014 May 3. PMID 24798886
- [Background] Rabin LA, Smart CM, Crane PK, Amariglio RE, Berman LM, Boada M, Buckley RF, Chetelat G, Dubois B, Ellis KA, Gifford KA, Jefferson AL, Jessen F, Katz MJ, Lipton RB, Luck T, Maruff P, Mielke MM, Molinuevo JL, Naeem F, Perrotin A, Petersen RC, Rami L, Reisberg B, Rentz DM, Riedel-Heller SG, Risacher SL, Rodriguez O, Sachdev PS, Saykin AJ, Slavin MJ, Snitz BE, Sperling RA, Tandetnik C, van der Flier WM, Wagner M, Wolfsgruber S, Sikkes SA. Subjective Cognitive Decline in Older Adults: An Overview of Self-Report Measures Used Across 19 International Research Studies. J Alzheimers Dis. 2015 Sep 24;48 Suppl 1(0 1):S63-86. doi: 10.3233/JAD-150154. PMID 26402085
- [Background] Reisberg B, Shulman MB, Torossian C, Leng L, Zhu W. Outcome over seven years of healthy adults with and without subjective cognitive impairment. Alzheimers Dement. 2010 Jan;6(1):11-24. doi: 10.1016/j.jalz.2009.10.002. PMID 20129317
- [Background] Amariglio RE, Mormino EC, Pietras AC, Marshall GA, Vannini P, Johnson KA, Sperling RA, Rentz DM. Subjective cognitive concerns, amyloid-beta, and neurodegeneration in clinically normal elderly. Neurology. 2015 Jul 7;85(1):56-62. doi: 10.1212/WNL.0000000000001712. Epub 2015 Jun 5. PMID 26048028
- [Background] Mecocci P, Tinarelli C, Schulz RJ, Polidori MC. Nutraceuticals in cognitive impairment and Alzheimer's disease. Front Pharmacol. 2014 Jun 23;5:147. doi: 10.3389/fphar.2014.00147. eCollection 2014. PMID 25002849
- [Background] Okuyama S, Morita M, Kaji M, Amakura Y, Yoshimura M, Shimamoto K, Ookido Y, Nakajima M, Furukawa Y. Auraptene Acts as an Anti-Inflammatory Agent in the Mouse Brain. Molecules. 2015 Nov 10;20(11):20230-9. doi: 10.3390/molecules201119691. PMID 26569206
- [Background] Okuyama S, Kanzaki T, Kotani Y, Katoh M, Sawamoto A, Nakajima M, Furukawa Y. Continual Treatment with the Peels of Citrus kawachiensis (Kawachi Bankan) Protects against Dopaminergic Neuronal Cell Death in a Lipopolysaccharide-Induced Model of Parkinson's Disease. J Nutr Sci Vitaminol (Tokyo). 2019;65(2):205-208. doi: 10.3177/jnsv.65.205. PMID 31061292
- [Background] Ghofrani S, Joghataei MT, Mohseni S, Baluchnejadmojarad T, Bagheri M, Khamse S, Roghani M. Naringenin improves learning and memory in an Alzheimer's disease rat model: Insights into the underlying mechanisms. Eur J Pharmacol. 2015 Oct 5;764:195-201. doi: 10.1016/j.ejphar.2015.07.001. Epub 2015 Jul 3. PMID 26148826
- [Background] Okuyama S, Kotani Y, Yamamoto K, Sawamoto A, Sugawara K, Sudo M, Ohkubo Y, Tamanaha A, Nakajima M, Furukawa Y. The peel of Citrus kawachiensis (kawachi bankan) ameliorates microglial activation, tau hyper-phosphorylation, and suppression of neurogenesis in the hippocampus of senescence-accelerated mice. Biosci Biotechnol Biochem. 2018 May;82(5):869-878. doi: 10.1080/09168451.2018.1433993. Epub 2018 Feb 9. PMID 29424280
- [Background] Sanchez-Rodriguez E, Biel-Glesson S, Fernandez-Navarro JR, Calleja MA, Espejo-Calvo JA, Gil-Extremera B, de la Torre R, Fito M, Covas MI, Vilchez P, Alche JD, Martinez de Victoria E, Gil A, Mesa MD. Effects of Virgin Olive Oils Differing in Their Bioactive Compound Contents on Biomarkers of Oxidative Stress and Inflammation in Healthy Adults: A Randomized Double-Blind Controlled Trial. Nutrients. 2019 Mar 6;11(3):561. doi: 10.3390/nu11030561. PMID 30845690
- [Background] ThyagaRajan S, Priyanka HP. Bidirectional communication between the neuroendocrine system and the immune system: relevance to health and diseases. Ann Neurosci. 2012 Jan;19(1):40-6. doi: 10.5214/ans.0972.7531.180410. PMID 25205962
- [Derived] Rolandi E, Dodich A, Mandelli S, Canessa N, Ferrari C, Ribaldi F, Munaretto G, Ambrosi C, Gasparotti R, Violi D, Iannaccone S, Marcone A, Falini A, Frisoni GB, Galluzzi S, Cerami C, Cavedo E. Targeting brain health in subjective cognitive decline: insights from a multidomain randomized controlled trial. Aging Clin Exp Res. 2025 May 14;37(1):151. doi: 10.1007/s40520-025-03062-z. PMID 40366507
- [Derived] Galluzzi S, Marizzoni M, Gatti E, Bonfiglio NS, Cattaneo A, Epifano F, Frisoni GB, Genovese S, Geviti A, Marchetti L, Sgro G, Solorzano CS, Pievani M, Fiorito S. Citrus supplementation in subjective cognitive decline: results of a 36-week, randomized, placebo-controlled trial. Nutr J. 2024 Nov 1;23(1):135. doi: 10.1186/s12937-024-01039-8. PMID 39482712
- [Derived] Galluzzi S, Zanardini R, Ferrari C, Gipponi S, Passeggia I, Rampini M, Sgro G, Genovese S, Fiorito S, Palumbo L, Pievani M, Frisoni GB, Epifano F. Cognitive and biological effects of citrus phytochemicals in subjective cognitive decline: a 36-week, randomized, placebo-controlled trial. Nutr J. 2022 Oct 17;21(1):64. doi: 10.1186/s12937-022-00817-6. PMID 36253765
- See also: Related Info — https://www.elsevier.com/books/the-neuroendocrine-immune-network-in-ageing/straub/978-0-444-51617-6